CLINICAL TRIAL: NCT05628779
Title: Evaluation of the Safety, Efficacy and Cost-effectiveness of Transcatheter Tricuspid Valve Repair in Patients With Severe Tricuspid Regurgitation in the Netherlands.
Brief Title: Evaluating Edge-to-edge Transcatheter Tricuspid Valve Repair in Patients With Severe Symptomatic Tricuspid Regurgitation
Acronym: TRACE-NL
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Martin J. Swaans, Principal Investigator, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL81645.100.22
Record Dates: First submitted 2022-10-27; First posted 2022-11-29 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Tricuspid Valve Regurgitation, Nonrheumatic; Cardiac Catheterization; Heart Failure, Right Sided; Valve Regurgitation, Tricuspid
Keywords: Transcatheter tricuspid valve repair; Tricuspid valve regurgitation; Tricuspid valve; Leaflet approximation devices
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Failure

STUDY DESIGN:
Intervention Model Description: A total of 150 patients will be randomly assigned with a 2:1 allocation to either interventional (n=100) or control group (n=50).
Masking Description: Randomized controlled trial with open-label extension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Transcatheter Edge-to-Edge Repair (TEER) on top of the Standard Of Care (SOC) (Experimental): Transcatheter Edge-to-Edge Repair (TEER) on top of the Standard Of Care (SOC)
  Interventions: Device: TriClip TTVr system (Abbott Vascular); Device: PASCAL TTVr system (Edwards Lifesciences)
- Standard Of Care (SOC) (No Intervention): Patients will continue the SOC with heart failure medication following the European Society of Cardiology guideline 2021 recommendations (e.g. diuretics)

INTERVENTIONS:
Device: TriClip TTVr system (Abbott Vascular) — Edge-to-edge leaflet approximation for the tricuspid valve
  Arms: Transcatheter Edge-to-Edge Repair (TEER) on top of the Standard Of Care (SOC)
Device: PASCAL TTVr system (Edwards Lifesciences) — Edge-to-edge leaflet approximation for the tricuspid valve
  Arms: Transcatheter Edge-to-Edge Repair (TEER) on top of the Standard Of Care (SOC)

SUMMARY:
This is a national multicenter, open-label, randomized controlled trial to show superiority of edge-to-edge Transcatheter Tricuspid Valve repair (TTVr) on top of the Standard Of Care (SOC; heart failure medication) over the SOC alone in patients with symptomatic severe Tricuspid Regurgitation (TR) in the Netherlands.

DETAILED DESCRIPTION:
Tricuspid valve regurgitation (TR) is a common heart valve disease associated with mortality, heart failure hospitalization (HHF) and a significant negative impact on quality of life (QoL). The prevalence of moderate or severe TR in the Netherlands is estimated at 0.55% and becoming more prevalent. Surgery is rarely performed, because in-hospital mortality is high and there is little evidence for the efficacy. The majority of patients does therefore entirely dependent on treatment with heart failure medication. However, a subset of these patients experience (progressive) symptoms of refractory congestive heart failure despite the SOC with heart failure medication.

Transcatheter Tricuspid Valve repair (TTVr) offers several new strategies to address severe TR; one promising technique to treat patients with symptomatic severe TR is edge-to-edge tricuspid valve (TV) repair through leaflet approximation. Edge-to-edge TTVr may provide an elegant alternative treatment for many patients, because it is less burdensome due to the minimally invasive nature. Moreover, multiple single-arm trials already reported promising outcomes in terms of efficacy and safety, and the technique is very similar to Transcatheter Mitral Valve repair (TMVr), with yet proven feasibility, efficacy and safety.

The aim of this study is to evaluate the safety, efficacy and cost-effectiveness of TTVr for patients with symptomatic severe TR despite the SOC and high/prohibitive surgical risk in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is symptomatic (New York Heart Association Functional Class II, III or ambulatory class IV) despite Standard Of Care (SOC). The Central Screening Committee (CSC) will assess whether the patient is receiving SOC. The CSC will also ensure that in case of the presence of atrial fibrillation, left sided heart valve disease (not requiring intervention) or coronary artery disease, conditions are first treated adequately with medication and/or (surgical) intervention.
2. The patient suffers from ≥ grade 3 isolated TR as determined by the assessment of a qualifying transthoracic echocardiogram (TTE) and three-dimensional transesophageal echocardiogram (3DTEE) and confirmed by the CSC, according to European Association for Percutaneous Cardiovascular Interventions (Tricuspid Focus Group) consensus document (in press). Note: If cardiac procedure(s) occur after eligibility was determined, TR grade will be re-assessed 30 days after the procedure.
3. The cardiac surgeon of the sites' local heart team concurs that the patient is at high estimated risk for mortality or morbidity with TV surgery.
4. The patient is ≥18 years of age at time of consent.
5. The patient must provide written informed consent prior to any trial related procedure.

Exclusion Criteria:

1. Systolic pulmonary artery pressure (sPAP) > 70 mmHg or fixed pre-capillary pulmonary hypertension as assessed by right heart catheterization. Severe uncontrolled hypertension Systolic Blood Pressure (SBP) ≥ 180 mmHg and/or Diastolic Blood Pressure (DBP) ≥ 110 mmHg.
2. Any condition that would interfere with a TTVr procedure, such as prior tricuspid valve repair or tricuspid valve leaflet anatomy which may preclude device implantation (e.g. calcification in grasping area, a severe coaptation defect of the tricuspid leaflets (no clip placement possible), pacemaker or Implantable Cardioverter Defibrillator (ICD) leads that would prevent appropriate placement or visualization of TTVr devices, Ebstein Anomaly (normal annulus position, but valve leaflets attached to walls and septum of the right ventricle), tricuspid valve anatomy non evaluable by echo, known allergy or hypersensitivity to dual antiplatelet therapy AND anticoagulant therapy or to device materials, femoral venous mass or thrombus or vegetation.
3. Indication for left-sided (e.g. severe aortic stenosis, severe mitral regurgitation) or pulmonary valve correction within prior 60 days. Note: concomitant mitral valve disease (e.g. mitral regurgitation) will be treated first and patients will be reassessed for the trial after 60 days.
4. Tricuspid valve stenosis - Defined as a tricuspid valve orifice of ≤ 1.0 cm2 and/or mean gradient ≥5 mmHg.
5. Left Ventricular Ejection Fraction (LVEF) ≤20%
6. Active endocarditis, active rheumatic heart disease, other ongoing infection requiring antibiotic therapy (enrolment possible 30 days after discontinuation of antibiotics with no active infection) or leaflets degenerated from rheumatic disease (i.e. noncompliant, perforated)
7. Myocardial infarction known unstable angina, or percutaneous coronary intervention within prior 30 days.
8. Hemodynamic instability defined as systemic systolic pressure <90 mmHg with or without afterload reduction, cardiogenic shock or the need for inotropic support or hemodynamic support device (e.g. intra-aortic balloon pump).
9. Cerebrovascular Accident (CVA) within prior 90 days
10. Chronic dialysis
11. Bleeding disorders or hypercoagulable state, inability to use dual antithrombotic therapy due to contraindication, allergy or hypersensitivity
12. Active peptic ulcer or active gastrointestinal (GI) bleeding
13. Life expectancy of less than 12 months
14. Subject currently participating in another clinical trial (not yet completed primary endpoint) or in another clinical investigation for valvular heart disease.
15. Pregnant or nursing patients or those who plan pregnancy during the course of the trial. Women of childbearing age are required to have a negative pregnancy test 7 days prior to baseline visit. Women of childbearing age should be instructed to use safe contraception or have a sterilized regular partner.
16. Presence of anatomic or comorbid conditions, or other medical, social or psychological conditions that, in the eye of the investigator, limits the subject's ability to participate in the clinical investigation or comply with follow-up requirements, or impact the scientific soundness of the investigation results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite of all-cause mortality, heart failure hospitalization and Quality of Life | 12 months
  Quality of Life is measured with the Kansas City Cardiomyopathy Questionnaire with a 5 point change as clinically significant (0-100 points, higher score is better outcome)

SECONDARY OUTCOMES:
All-cause mortality | 12 months
  Mortality of any cause
Hospitalization for heart failure | 12 months
  Hospitalization for acute decompensated heart failure
Change in Kansas City Cardiomyopathy Questionnaire | 12 months
  5 point change is considered clinically significant (0-100 points with higher score is a better outcome), change of 5 points in Kansas City Cardiomyopathy Questionnaire is considered clinically meaningful
Number of participants without Major Adverse Events (MAE) | 30 days and 12 months
  Cardiovascular mortality, myocardial infarction, stroke, major bleeding, device embolisation, new onset renal failure, endocarditis requiring surgery, non-elective cardiovascular surgery for device related adverse events.
Change in New York Heart Association | 12 months
  ranging from 0 to 4 (no limitation to severe limitation)
Change in 6-Minute Walk Test | 12 months
  Distance in meters (higher score is a better outcome)
Reduction tricuspid regurgitation | 30 days, 6 months and 12 months
  Echocardiographic assessment of Tricuspid Regurgitation (at least from severe to moderate or less)
Cost-effectiveness as assessed by the Markov model | 12 months
  The investigators will compare the cost-effectiveness of the intervention group versus the control group based on lifetime horizon by constructing a Markov model with model parameters populated from the trial results as well as other published literature. The model will estimate the incremental cost-effectiveness ratio between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: M.J. Swaans, MD,PhD, Principal Investigator — St. Antonius Hospital
Locations (6):
- Netherlands (6):
  - Amsterdam UMC, Amsterdam
  - UMC Groningen, Groningen
  - Leiden UMC, Leiden
  - Maastricht UMC+, Maastricht
  - St. Antonius Hospital Nieuwegein, Nieuwegein
  - Erasmus University Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, the data will be locally saved at the st. Antonius Hospital and can be made available at request for reuse in other studies.
Supporting Information: Study Protocol, SAP
Time Frame: After publishing the main study articles, raw and modified data can be made available at request
Access Criteria: These criteria will be made in consultation with the legal advisor of our institution and have not yet been drafted.
  Specific degrees in the field of research have to be demonstrated, as wel as links with hospitals or research institutes of the researcher/physician (e.g. an employee contract)